CLINICAL TRIAL: NCT00925379
Title: Renal HYPODYSPLASIA;Study of Familial Cases and Search for Predisposing Genes
Brief Title: Renal HYPODYSPLASIA : Genetic and Familial Assessment
Acronym: HDR
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: P070151
Record Dates: First submitted 2009-06-19; First posted 2009-06-22 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: Renal HYPODYSPLASIA, Nonsyndromic, 1
MeSH Terms: conditions — Renal Hypodysplasia, Nonsyndromic, 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — DNA collection from the propositus and its parents and in case of families with more than one affected member, collection of DNA from the all family.
Oversight: Data Monitoring Committee: No

SUMMARY:
Evaluation of the frequency of familial cases of renal HYPODYSPLASIA

DETAILED DESCRIPTION:
DNA collection from the propositus and its family. A questionnaire will be filled by the parents to seek other affected individual in the family.With another affected member, DNA collection will be collected from the whole family.

A renal ultrasound will be prescribed for the parents, brothers and sisters.

ELIGIBILITY:
Inclusion criteria :

- Children aged more than 3 months and less than 18 years old with a renal bilateral HYPODYSPLASIA set by renal ultrasound examination :

* renal size < -2DS
* with/or hyperechogenicity or lack of cortical-medullary differentiation
* with/or renal cysts

Exclusion criteria :

* Bladder uropathy or sus-bladder uropathy
* Recessive or dominant renal polycystic disease
* Bardet-Biedl syndrome and other malformative syndromes except renal coloboma syndrome, Renal cysts and diabetes syndrome RCAD
* Lack of written informed consent

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with a bilateral renal hypodysplasia
Sampling Method: Non-Probability Sample
Enrollment: 342 (Actual)
Dates: Start 2009-04; Primary Completion 2013-04 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Evaluation of the heritability of renal HYPODYSPLASIA (on the renal ultra sound) and DNA collection to make possible identification of predisposing genes | the same day

CONTACTS AND LOCATIONS:
Overall Officials: Remi Salomon, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Vincent Guigonis, MD, PhD, Principal Investigator — University Hospital, Limoges
Locations (1):
- Necker Hospital, Paris, France